CLINICAL TRIAL: NCT03888807
Title: The Effect of Biofreeze® vs. a Placebo on Knee Osteoarthritis Walking Gait Characteristics and Pain
Brief Title: Biofreeze® vs. a Placebo on Knee Osteoarthritis Walking Gait Characteristics and Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Decided not go move forward with this population as recruitment was difficult
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BFvP KneeOA Walking
Record Dates: First submitted 2018-07-02; First posted 2019-03-25 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Topical Analgesic
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 1 of 2 topicals, Gel A or Gel B. Upon completion of study procedures they will return for a second testing session and receive the other topical.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, and statistician will be blind to the intervention received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofreeze (Experimental): The Biofreeze® gel will contain 3.5% menthol while the placebo will be the same formula with menthol removed and a menthol fragrance added so it is non-distinguishable from the real Biofreeze® gel. The dose of both gels will be 5 mL per knee, which is consistent with previous studies who reported a treatment effect for topical gels containing menthol (1 mL of gel for every 200 cm2 of surface area). The treatment will be applied by the investigator using a gloved hand and syringe containing 5mL of gel. The gel will be applied to the anterior and posterior knee from superior patella to the quadriceps insertion over a period of 5 seconds. The participant will wait 15 minutes, rate the pain in their knees.
  Interventions: Drug: Biofreeze
- Placebo (Sham Comparator): The Biofreeze® gel will contain 3.5% menthol while the placebo will be the same formula with menthol removed and a menthol fragrance added so it is non-distinguishable from the real Biofreeze® gel. The dose of both gels will be 5 mL per knee, which is consistent with previous studies who reported a treatment effect for topical gels containing menthol (1 mL of gel for every 200 cm2 of surface area). The treatment will be applied by the investigator using a gloved hand and syringe containing 5mL of gel. The gel will be applied to the anterior and posterior knee from superior patella to the quadriceps insertion over a period of 5 seconds. The participant will wait 15 minutes, rate the pain in their knees
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Biofreeze — Biofreeze is a topical analgesic that uses the cooling effect of menthol, a natural pain reliever, to soothe minor muscle and joint pain. The product will be applied immediately after walking. The participant will wait 15 minutes prior to walking again.
  Arms: Biofreeze
Drug: Placebo — The placebo is the Biofreeze product with all active ingredients removed. The product will be applied immediately after walking. The participant will wait 15 minutes prior to walking again.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of Biofreeze® versus a placebo on walking gait characteristics and pain during walking in individuals with bilateral knee osteoarthritis (OA).

DETAILED DESCRIPTION:
A convenience sample of 20 participants, >40 years with previously diagnosed bilateral KOA were recruited. Participants must have been diagnosed with bilateral knee OA and be able to perform all study procedures. All participants reported in comfortable clothing and sneakers. After explanation of the study and consent, participants completed the demographics questionnaire, Numeric Pain Rating Scale (NPRS), Western Ontario and McMaster Universities Arthritis Index (WOMAC), and knee function survey. Participants then completed a 3mph 3-minute walking baseline assessment. Following the assessment, participants rated their pain and were randomly assigned to receive a blinded topical of either Biofreeze® or a Placebo. The dose of both gels was 5 mL per knee. The participant then waited 15 minutes, rated their pain, and repeated the 3-minute walking assessment and rated their pain once more. There was a minimum of a 24-72-hour washout period after which time the participants repeated the same protocol using the other topical.

ELIGIBILITY:
Inclusion Criteria:

* must have been diagnosed with bilateral knee osteoarthritis (OA) and be able to perform all study procedures

Exclusion Criteria:

* less than 40 years of age, pregnancy, cancer, rheumatoid arthritis, a total or partial knee replacement, and/or a corticosteroid injection within the past 4 weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale | Pain will be measured at baseline, immediately following the 3 minute walk, 15 minutes after topical application, and after the second 3 minute walk for both topical applications
  Pain will be measures on a scale of 0 to 10, 0 being no pain at all and 10 representing the worst imaginable pain.
Change in Knee Flexion | Knee Flexion Range of Motion will be measured for both topical applications at initial walk and post-topical walk. The session will last a total of 30 minutes.
  Knee Flexion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera and will be measured during the last 30 seconds of the 3 minute walk.
Change inHip Flexion | Knee Flexion Range of Motion will be measured for both topical applications at initial walk and post-topical walk. The session will last a total of 30 minutes
  Hip Flexion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera and will be measured during the last 30 seconds of the 3 minute walk.
Change in Step Length | Knee Flexion Range of Motion will be measured for both topical applications at initial walk and post-topical walk. The session will last a total of 30 minutes
  Step Length will be measured using the Woodway Walker View Treadmill which utilizes load cells within the treadmill belt and will be measured during the last 30 seconds of the 3 minute walk.

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No